CLINICAL TRIAL: NCT02178202
Title: Prescription of Two Exercise Therapy Protocols for Treating Chronic Low Back Pain
Brief Title: McKenzie Exercise Vs Harmonic Technique in Chronic Low Back Pain
Acronym: CLBP
Status: No longer available | Type: Expanded Access
Sponsor: University of Tehran (Other)
Responsible Party: Principal Investigator, Rahman Sheikhhoseini, PHD candidates, University of Tehran
Other Study IDs: qs-2012-05-05
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Low Back Pain
Keywords: Harmonic technique, Low Back Pain, McKenzie exercise, Pain, Disability
MeSH Terms: conditions — Low Back Pain; Pain

INTERVENTIONS:
Behavioral: McKenzie exercise — First to sixth McKenzie exercises were performed for 5 times/week and 10 treatment sessions totally.
Device: Harmonic technique — Lower limb suspension exercise was performed for 5 times/week and 10 treatment sessions totally

SUMMARY:
The purpose of this study was to investigate the effects of HT compared with McK exercise on pain and disability in patients with LBP.

ELIGIBILITY:
Inclusion Criteria:

* Had persistent back pain at least eight weeks or during the last year subjects must suffer from LBP at least three times and each time lasted more than a week.

Exclusion Criteria:

* Had a history of fracture or surgery in the spine, pelvis and lower extremities through last year
* History of neuromuscular disease
* The referral and radicular pain in the lower extremities and neurological or sensory disturbance in the lower extremities
* Urinary incontinence and pain severity higher that 7 based on visual analogue scale (VAS)

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult